CLINICAL TRIAL: NCT02141269
Title: Comparative Effectiveness of Pocket, Mobile, Hand-held Echocardiography and Conventional Transthoracic Echocardiography in an Inpatient and Outpatient Clinical Setting
Brief Title: Comparitive Effectiveness of PME Versus Transthoracic Echocardiogram (TTE)
Status: Completed | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Principal Investigator, Eric Topol, MD, Principal Investigator, Scripps Translational Science Institute
Other Study IDs: 12-5906
Record Dates: First submitted 2012-06-28; First posted 2014-05-19 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Cardiac Disease
Keywords: Transthoracic echocardiogram; Hand-held Echocardiography
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A new hand held pocket echo device (GE Vscan) has now become available to clinicians, with limited data available comparing the effectiveness of this device as a screening tool when compared to traditional transthoracic echocardiography (TTE).

The investigators are evaluating the effectiveness of this hand-held echo (HHE) device in detecting cardiac pathology in a both an inpatient and outpatient clinical setting as compared to a comprehensive TTE evaluation.

DETAILED DESCRIPTION:
A new hand held pocket echo device (GE Vscan) has now become available to clinicians, with limited data available comparing the effectiveness of this device as a screening tool when compared to TTE.

We are evaluating the effectiveness of this HHE device in detecting cardiac pathology in a both an inpatient and outpatient clinical setting as compared to a comprehensive TTE evaluation.

This study compares the images from the two modalities with regards to multiple parameters typically evaluated by traditional TTE. This would include the following:

1. Ejection fraction: estimates how well the heart is squeezing/functioning.
2. Segmental wall motion abnormalities: if one wall of the heart is not moving well, this suggests that part of the heart is not getting enough blood supply and could represent a blockage in a blood vessel supplying the heart or in other terms a heart attack.
3. Left ventricular end-diastolic dimension: allows us to see if the heart is dilated
4. Inferior vena cava size: the size of this great vein can help estimate if patient has too much fluid in their vascular bed.
5. Aortic valve pathology: whether or not there is thickening of the valve or impairment of it's opening.
6. Mitral valve pathology: whether or not the valve is significantly thickened or with impaired closing and opening.
7. Pericardial effusion: excessive fluid in the sack around the heart.

The images obtained on the HHE will be evaluated by two experienced echocardiographers as well as two cardiology fellows who have obtained training in image acquisition and interpretation. The readers of the HHE images are blinded to the TTE results, and vice versa.

A comparison of these individual parameters on HHE and TTE allows us to validate this new, convenient screening tool in detecting cardiac pathology.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects with an order for a routine transthoracic echocardiogram based on clinical indications.
2. Vscan images will be obtained to evaluate multiple parameters (noted on research summary).
3. Immediately after Vscan imaging, a complete transthoracic echocardiogram will be performed.
4. Images will be compared between the Vscan device and the traditional transthoracic echocardiogram.

Exclusion Criteria:

1. Subjects who had a limited transthoracic echocardiography (i.e limited views)
2. Vscan imaging not attempted for a certain parameter

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inpatient and outpatient subjects with an order for a routine transthoracic echocardiogram based on clinical indications.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Comparison of HHE and TTE results | 1 time
  Comparison of the two modalities includes accuracy, sensitivity, specificity, proportion visualized, and inter-observer variability.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Topol, MD, Principal Investigator — Scripps Health
Locations (1):
- Scripps Green Hospital, La Jolla, California, United States